CLINICAL TRIAL: NCT05451810
Title: A Phase 2, Open-Label Trial to Evaluate Safety of Epcoritamab Monotherapy in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma and Classic Follicular Lymphoma (Previously Grade 1-3a) When Administered in the Outpatient Setting
Brief Title: A Study to Evaluate Adverse Events of Subcutaneous (SC) Epcoritamab Administered in the Outpatient Setting in Adult Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma and Classic Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-362
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-Cell Lymphoma; Classic Follicular Lymphoma
Keywords: Relapsed or Refractory Diffuse Large B-Cell Lymphoma; Relapsed or Refractory Classic Follicular Lymphoma; Non-Hodgkins Lymphoma; Cancer; Epcoritamab; ABBV-GMAB-3013; EPCORE
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Main Cohort: Epcoritamab Diffuse Large B-Cell Lymphoma (DLBCL) (Experimental): Participants with relapsed or refractory (R/R) DLBCL will receive subcutaneous (SC) epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab
- Main Cohort: Epcoritamab Classic Follicular Lymphoma (cFL) (Experimental): Participants with R/R cFL will receive SC epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab
- Diversity Enriched Cohort: Epcoritamab DLBCL (Experimental): Participants with R/R DLBCL will receive SC epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab
- Diversity Enriched Cohort: Epcoritamab cFL (Experimental): Participants with R/R cFL will receive SC epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection (SC)
  Other Names: ABBV-GMAB-3013

SUMMARY:
B-cell Lymphoma is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections). Classic Follicular Lymphoma is a slow-growing type of non-Hodgkin lymphoma. The purpose of this study is to assess the safety of epcoritamab in adult participants in relapsed or refractory (R/R) diffuse large b-cell lymphoma (DLBCL) who have received at least 1 prior line of systemic antilymphoma therapy including at least 1 anti-CD20 monoclonal antibody-containing therapy or R/R classic follicular lymphoma (cFL). Adverse events will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of R/R DLBCL and R/R cFL. Study doctors will assess participants in a monotherapy treatment arm of epcoritamab. Participants will receive escalating doses of epcoritamab, until full dose is achieved. Approximately 184 adult participants with R/R DLBCL and R/R cFL will be enrolled in the study in approximately 80 sites in the United States of America.

Participants will receive escalating doses of subcutaneous epcoritamab, until full dose is achieved, in 28-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy >3 months on standard of care (SOC) treatment.
* Meets the following disease activity criteria:

  -- Relapsed or Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL):
  * Documented CD20+ mature B-cell neoplasm according to the the 5th edition of World Health Organization (WHO) classification of Haematolymphoid Tumours, based on most recent representative pathology report;
  * Diffuse large B-cell lymphoma, not otherwise specified (NOS) (de novo or transformed from follicular lymphoma (FL) or Marginal Zone Lymphoma [MZL]);
  * High-grade B-cell Lymphoma including "double-hit" or "triple-hit" DLBCL (technically classified in WHO 2022 or 2016 as high-grade B-cell lymphoma [HGBCL], with MYC and BCL2 and/or BCL6 translocations).
  * Follicular large B-cell lymphoma (FLBL, formerly FL grade 3B);
  * Relapsed or refractory disease and previously treated with at least 1 prior systemic antineoplastic therapies including at least 1 anti-CD20 monoclonal antibody-containing therapy; Note: Relapsed disease is defined as disease that previously responded to therapy but progressed >= 6 months after completion of therapy. Refractory disease is defined as disease that either progressed during therapy, failed to achieve an objective response to prior therapy, or progressed within 6 months after completion of therapy (including maintenance therapy).
  * Either failed prior autologous hematopoietic stem cell transplantation (HSCT), or ineligible for autologous HSCT including but not limited to age, Eastern Cooperative Oncology Group (ECOG) performance status, participant decision, comorbidities and/or insufficient response to prior treatment.
* R/R Follicular Lymphoma:

  * Documented CD20+ mature B-cell neoplasm according to the 5th edition of WHO classification of Haematolymphoid Tumours, based on representative pathology report;

    --- Classic FL (cFL) (previously FL grade 1, 2, or 3a) without clinical or pathological evidence of transformation;
  * Relapsed or refractory disease and previously treated with at least 2 prior lines of systemic antineoplastic therapies including at least 1 anti-CD20 monoclonal antibody containing therapy; Note: Relapsed disease is defined as disease that previously responded to therapy but progressed >= 6 months after completion of therapy. Refractory disease is defined as disease that either progressed during therapy, failed to achieve an objective response to prior therapy, or progressed within 6 months after completion of therapy (including maintenance therapy).
  * Previously treated with an alkylating agent or lenalidomide;
  * Relapsed or refractory to the last prior line therapy. Previous lymphoma therapy is defined as 1 of the following: At least 2 months of single-agent therapy, at least 2 consecutive cycles of combination therapy, autologous HSCT, immunomodulatory therapy, or radioimmunotherapy.
* Has at least one target lesion defined as:

  * >= 1 measurable nodal lesion (long axis > 1.5 cm) and/or >= 1 measurable extranodal lesion (long axis > 1.0 cm) on CT (or MRI) AND
  * FDG PET scan demonstrating positive lesion(s) compatible with CT (or MRI) defined anatomical tumor sites.
* Must have ECOG performance status 0 - 2.
* Must have acceptable organ (renal, liver, and hematologic) function within the screening period prior to the first dose of study drug:

  * Absolute neutrophil count (ANC) >= 1.0 × 10^9/L (growth factor support allowed in case of bone marrow involvement, but participant must have not received growth factor within 14 days prior to screening lab collection);
  * Hemoglobin >= 8.0 g/dL (RBC transfusions permitted, but participants must not have received blood transfusions within 7 days prior to Screening lab collection);
  * Platelet count >= 75 × 10^9/L, or >= 50 × 10^9/L in the presence of bone marrow involvement or splenomegaly (platelet transfusions are permitted, but participants must not have received blood transfusions within 7 days prior to Screening lab collection);
  * International normalized ratio (INR) (or Prothrombin Time [PT]) and aPTT <= 1.5 × upper limit of normal (ULN), unless receiving anticoagulation
  * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) <= 3.0 × upper limit of normal (ULN); unless due to hepatic involvement of disease or non-hepatic origin. For participants with hepatic involvement of disease, serum AST and serum ALT <= 5.0 × ULN
  * Direct bilirubin <= 2 × ULN;
  * Estimated creatine clearance (CrCl) as calculated by Cockcroft-Gault Formula >= 45 mL/min, or estimated glomerular filtration rate (eGFR) as calculated by Modification of Diet in Renal Disease [MDRD] equation >= 45 mL/min;
  * Lymphocyte count < 5 × 10^9/L.

Exclusion Criteria:

* Have a primary central nervous system (CNS) lymphoma or known CNS involvement by lymphoma including leptomeningeal disease, at screening as confirmed by magnetic resonance imaging (MRI)/computed tomography (CT) scan (brain) and, if clinically indicated, by lumbar puncture.
* Uncontrolled Human Immunodeficiency Virus (HIV) infection. HIV viral load that is undetectable and controlled with medication for at least 1 year prior to enrollment is allowed. Note: If participant has no history of HIV infection, HIV testing does not need to be conducted at screening unless it is required per local guidelines or institutional standards.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Grade 3 or Higher Cytokine Release Syndrome (CRS) Events | Up to 3 Months
  Cytokine Release Syndrome events will be graded using American Society for Transplantation and Cellular Therapy (ASTCT), with a higher grade indicating higher severity.
Percentage of Participants Experiencing Grade 3 or Higher Immune Cell-Associated Neurotoxicity Syndrome (ICANS) Events | Up to 3 Months
  ICANS events will be graded using ASTCT, with a higher grade indicating higher severity.
Percentage of Participants Experiencing Grade 3 or Higher Neurotoxicity (Ntox) Events | Up to 3 Months
  Ntox is defined as the percentage of participants who developed at least 1 Grade 3 or higher Ntox since the initiation of epcoritamab treatment.

SECONDARY OUTCOMES:
Best Overall Response (BOR) Determined by Lugano 2014 Criteria Per Investigator Assessment | Up to 3 Months
  BOR is defined as the percentage of participants who achieved best overall response of complete response (CR) or partial response (PR) determined by Lugano 2014 criteria as assessed by investigators.
CR Determined by Lugano 2014 Criteria Per Investigator Assessment | Up to 3 Months
  Complete response is defined as the percentage of participants who achieved best overall response of CR determined by Lugano 2014 criteria as assessed by investigator.
Diversity Enriched Cohort: Incidence of Treatment-Emergent Adverse Events (TEAEs) by Severity Level | Up to 3 Months
  Treatment-emergent events (TEAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Diversity Enriched Cohort: Severity of TEAEs by Severity Level | Up to 3 Months
  Treatment-emergent events (TEAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Diversity Enriched Cohort: Incidence of Serious Adverse Events (SAEs) by Severity Level | Up to 3 Months
  A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Diversity Enriched Cohort: Severity of SAEs by Severity Level | Up to 3 Months
  A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Diversity Enriched Cohort: Median Time to Onset of CRS of Grade 3 or Higher | Up to 3 Months
  Median time to onset of CRS of Grade 3 or higher.
Diversity Enriched Cohort: Median Time to Resolution of CRS of Grade 3 or Higher | Up to 3 Months
  Median time to resolution of CRS of Grade 3 or higher.
Diversity Enriched Cohort: Median Time to Onset of ICANS of Grade 3 or Higher | Up to 3 Months
  Median time to onset of ICANS of Grade 3 or higher.
Diversity Enriched Cohort: Median Time to Resolution of ICANS of Grade 3 or Higher | Up to 3 Months
  Median time to resolution of ICANS of Grade 3 or higher.
Diversity Enriched Cohort: Median Time to Onset of Ntox of Grade 3 or Higher | Up to 3 Months
  Median time to onset of Ntox of Grade 3 or higher.
Diversity Enriched Cohort: Median Time to Resolution of Ntox of Grade 3 or Higher | Up to 3 Months
  Median time to resolution of Ntox of Grade 3 or higher.
Diversity Enriched Cohort: Percentage of Participants Experiencing Any Adverse Events (AE)s | Up to 3 Months
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Diversity Enriched Cohort: Percentage of Participants Receiving Various Interventions for the Management of CRS After the First Full Dose of Epcoritamab | Up to 3 Months
  Percentage of participants receiving various interventions for the management of CRS after the first full dose of epcoritamab.
Diversity Enriched Cohort: Percentage of Participants Receiving Various Interventions for the Management of ICANS After the First Full Dose of Epcoritamab | Up to 3 Months
  Percentage of participants receiving various interventions for the management of ICANS after the first full dose of epcoritamab.
Diversity Enriched Cohort: Percentage of Participants Receiving Various Interventions for the Management of Ntox After the First Full Dose of Epcoritamab | Up to 3 Months
  Percentage of participants receiving various interventions for the management of Ntox after the first full dose of epcoritamab.
Diversity Enriched Cohort: Duration of response (DOR) | Up to 3 Months
  Duration of response is defined for participants who achieved BOR of CR or PR ('responders'), as the time in months from initial CR/PR to the earliest occurrence of disease progression determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Diversity Enriched Cohort: Progression-free survival (PFS) | Up to 3 Months
  Progression-free survival is defined as the time in months from the first dose of study drug to the earliest occurrence of disease progression determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Diversity Enriched Cohort: Overall survival (OS) | Up to 3 Months
  Overall survival is defined for as the time in months from first dose of epcoritamab to death from any cause.
Diversity Enriched Cohort: Time-to-response (TTR) | Up to 3 Months
  Time to response is defined for participants who achieved BOR of CR or PR ('responders') determined by Lugano 2014 criteria as assessed by investigator, as the time in months from first dose of study drug to initial CR/PR.
Diversity Enriched Cohort: Duration of CR (DOCR) | Up to 3 Months
  The duration of complete response is defined for participants who achieved BOR of CR (Complete Responders), as the duration from the first CR response to the earliest date of disease progression determined per Lugano 2014 criteria, as assessed by the investigator, or death, whichever occurs first.
Diversity Enriched Cohort: Time to Next Treatment | Up to 3 Months
  Time to next treatment is defined as the time from the date of the first dose of study drug to the start of new non-protocol-specified treatment or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (72):
- United States (70):
  - Infirmary Health - Infirmary Cancer Care at Mobile Infirmary /ID# 264630, Mobile, Alabama
  - University of Arkansas for Medical Sciences /ID# 244562, Little Rock, Arkansas
  - Highlands Oncology Group, PA /ID# 245002, Springdale, Arkansas
  - Beverly Hills Cancer Center /ID# 255327, Beverly Hills, California
  - Compassionate Cancer Care Research Group - Fountain Valley /ID# 246133, Fountain Valley, California
  - UCSF Fresno /ID# 263286, Fresno, California
  - University of California, Los Angeles /ID# 244573, Los Angeles, California
  - Rocky Mountain Cancer Centers - Boulder /ID# 247653, Boulder, Colorado
  - Bennett Cancer Center - Stamford Hospital /ID# 244530, Stamford, Connecticut
  - MedStar Washington Hospital Center /ID# 246068, Washington D.C., District of Columbia
  - Cancer Specialists of North Florida /ID# 261842, Jacksonville, Florida
  - Florida Cancer Specialists /ID# 260854, Lake Mary, Florida
  - Mount Sinai Medical Center-Miami Beach /ID# 249045, Miami Beach, Florida
  - Memorial Hospital West /ID# 248432, Pembroke Pines, Florida
  - BRCR Medical Center Inc /ID# 262527, Tamarac, Florida
  - Cleveland Clinic Florida /ID# 244532, Weston, Florida
  - Emory University, Winship Cancer Institute /ID# 246056, Atlanta, Georgia
  - University of Illinois at Chicago /ID# 245038, Chicago, Illinois
  - Illinois Cancer Specialists /ID# 247655, Niles, Illinois
  - Parkview Comprehensive Cancer Center /ID# 244545, Fort Wayne, Indiana
  - Indiana Blood & Marrow Transpl /ID# 244971, Indianapolis, Indiana
  - University of Iowa Health Care /ID# 258227, Des Moines, Iowa
  - Our Lady Of The Lake Regional Medical Center /ID# 255008, Baton Rouge, Louisiana
  - American Oncology Partners of Maryland /ID# 244968, Bethesda, Maryland
  - Maryland Oncology Hematology /ID# 254192, Columbia, Maryland
  - Tufts Medical Center /ID# 246074, Boston, Massachusetts
  - Massachusetts General Hospital /ID# 245239, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 248651, Boston, Massachusetts
  - Cancer & Hematology Centers of Western Michigan - East /ID# 244985, Grand Rapids, Michigan
  - Trinity Health St. Joseph Mercy Ann Arbor /ID# 244547, Ypsilanti, Michigan
  - Hattiesburg Clinic /ID# 244980, Hattiesburg, Mississippi
  - St. Luke's Hospital - Chesterfield /ID# 247815, Chesterfield, Missouri
  - NHO - Nebraska Hematology-Oncology /ID# 263164, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center - 1 Medical Center Drive /ID# 245003, Lebanon, New Hampshire
  - The John Theurer Cancer /ID# 262532, Hackensack, New Jersey
  - Morristown Medical Center /ID# 244973, Morristown, New Jersey
  - University of New Mexico /ID# 252434, Albuquerque, New Mexico
  - New York Cancer & Blood Specialists - Lake Success Medical Oncology /ID# 264681, New Hyde Park, New York
  - Stony Brook University Medical Center /ID# 244631, New York, New York
  - New York Cancer and Blood Specialists - New York /ID# 264676, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 258610, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 244628, New York, New York
  - New York Cancer and Blood Specialists /ID# 259016, Port Jefferson Station, New York
  - New York Cancer and Blood Specialists - Bronx /ID# 264690, The Bronx, New York
  - East Carolina University - Brody School of Medicine /ID# 248989, Greenville, North Carolina
  - Wake Forest Univ HS /ID# 245005, Winston-Salem, North Carolina
  - Oncology Hematology Care, Inc. /ID# 246182, Cincinnati, Ohio
  - OhioHealth Arthur G.H. Bing, MD Cancer Center /ID# 260803, Columbus, Ohio
  - Toledo Clinic Cancer Center - Main /ID# 246852, Toledo, Ohio
  - University of Oklahoma, Stephenson Cancer Center /ID# 244568, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center /ID# 246410, Eugene, Oregon
  - Oregon Oncology Specialists in Salem /ID# 260570, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest /ID# 244984, Allentown, Pennsylvania
  - Spoknwrd Clinical Trials /ID# 265232, Easton, Pennsylvania
  - Penn State Milton S. Hershey Medical Center /ID# 244979, Hershey, Pennsylvania
  - UPMC Hillman Cancer Ctr /ID# 244571, Pittsburgh, Pennsylvania
  - Reading Hospital; McGlinn Cancer Institute /ID# 259181, West Reading, Pennsylvania
  - Prisma Health /ID# 247654, Greenville, South Carolina
  - The West Clinic /ID# 245004, Memphis, Tennessee
  - Vanderbilt University Medical Center /ID# 260953, Nashville, Tennessee
  - Texas Oncology - Austin Midtown /ID# 247656, Austin, Texas
  - Texas Oncology-Presbyterian Cancer Center Dallas /ID# 262659, Dallas, Texas
  - Texas Oncology - Dallas - Worth Street /ID# 262956, Dallas, Texas
  - University of Texas Southwestern Medical Center /ID# 244552, Dallas, Texas
  - Texas Oncology - San Antonio Medical Center /ID# 247658, San Antonio, Texas
  - Texas Oncology - Northeast Texas /ID# 247657, Tyler, Texas
  - Virginia Cancer Specialists - Gainesville /ID# 248760, Gainesville, Virginia
  - Virginia Oncology Associates - Norfolk (Lake Wright) /ID# 265514, Norfolk, Virginia
  - Blue Ridge Cancer Center /ID# 260597, Roanoke, Virginia
  - Northwest Medical Specialties - Tacoma /ID# 245045, Tacoma, Washington
- Puerto Rico (2):
  - Pan American Center for Oncology Trials, LLC /ID# 254952, Rio Piedras
  - Auxilio Mutuo Cancer Center /ID# 254953, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=M23-362